CLINICAL TRIAL: NCT02091128
Title: Pregnancy Chances in Classic Galactosemia
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: METC 13-4-127
Record Dates: First submitted 2014-03-13; First posted 2014-03-19 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Galactosemias; Primary Ovarian Insufficiency
MeSH Terms: conditions — Galactosemias; Primary Ovarian Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Females with classic galactosemia and POI

SUMMARY:
With this study, in which the incidence of pregnancy in classic galactosemia patients is studied, we aim to provide new insights to improve counselling. Our hypothesis is that the chance that a galactosemic woman with POI becomes pregnant is higher than the 5-10% that has been reported for women with POI due to other causes. Chance of spontaneous pregnancy will be evaluated through semi standardized interview in women with classic galactosemia aged 18 years or older. During the interview, questions will be asked regarding fertility and pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Classic galactosemia diagnosed by GALT enzyme activity assay or GALT-gene mutation analysis
* Eighteen years of age or older
* Diagnosed with POI defined as symptoms of hypergonadotrophic hypogonadism measured by serum concentrations of FSH and estradiol
* Capable of giving informed consent

Exclusion Criteria:

* Any known congenital or acquired disease or disorder negatively affecting pubertal development and/or fertility.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Academic hospital
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2014-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Pregnancy incidence despite POI diagnosis | day 1
  Will be assessed during semi-standardized interview

SECONDARY OUTCOMES:
Whether women have tried to conceive | day 1
  Will be assessed during semi-standardized interview
Time to pregnancy (in case a participant has been pregnant) | day 1
  Will be assessed during semi-standardized interview
Menstrual history | day 1
  Will be assessed during semi-standardized interview
Hormonal replacement therapy usage | day 1
  Will be assessed during semi-standardized interview

CONTACTS AND LOCATIONS:
Overall Officials: M. Estela Rubio-Gozalbo, Dr, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands

REFERENCES:
- [Background] Gubbels CS, Land JA, Rubio-Gozalbo ME. Fertility and impact of pregnancies on the mother and child in classic galactosemia. Obstet Gynecol Surv. 2008 May;63(5):334-43. doi: 10.1097/OGX.0b013e31816ff6c5. PMID 18419833